CLINICAL TRIAL: NCT04084548
Title: Lidocaine and Ketamine in Abdominal Surgery
Brief Title: Perioperative Lidocaine and Ketamine in Abdominal Surgery
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FLA 18-088
Record Dates: First submitted 2019-02-05; First posted 2019-09-10 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Pain
Keywords: Multimodal analgesia; Lidocaine; Ketamine; Abdominal surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine; Ketamine

STUDY DESIGN:
Intervention Model Description: Double-blind factorial randomization to lidocaine or placebo and ketamine or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Pharmacy-prepared medications.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Lidocaine and placebo (Experimental): Lidocaine and placebo
  Interventions: Drug: Lidocaine
- Ketamine and placebo (Experimental): Ketamine and placebo
  Interventions: Drug: Ketamine
- Lidocaine and ketamine (Experimental): Lidocaine and ketamine
  Interventions: Drug: Lidocaine and ketamine
- Placebo and placebo (Placebo Comparator): Placebo and placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine and ketamine — Perioperative lidocaine and ketamine infusion (see below for dosages and timings)
  Arms: Lidocaine and ketamine
Drug: Lidocaine — Perioperative lidocaine infusion (1.5 mg/kg bolus followed by an infusion of 2 mg/kg/hour based on actual body weight; the bolus and infusion will be started after anesthesia induction and before surgical incision, and continued until 1 hour after transfer from the operating room to the PACU)
  Arms: Lidocaine and placebo
Drug: Ketamine — Perioperative ketamine infusion (0.5 mg/kg bolus followed by an infusion of 0.3 mg/kg/hour based on actual body weight; the bolus and infusion will be started after anesthesia induction and before surgical incision, and continued until 1 hour after transfer from the operating room to the PACU)
  Arms: Ketamine and placebo
Drug: Placebo — Perioperative placebo infusion (normal saline)
  Arms: Placebo and placebo

SUMMARY:
The investigators propose to test the hypothesis that perioperative infusions of lidocaine and/or ketamine reduce opioid consumption and pain scores in adults recovering from elective inpatient abdominal surgery.

DETAILED DESCRIPTION:
The investigators propose a prospective, randomized, double-blind, placebo-controlled clinical trial (RCT) with a factorial design. Adults 18 to 80 years old having elective inpatient open or laparoscopic abdominal surgery with general anesthesia lasting 2 hours or longer will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 to 80 years old
* Elective inpatient open or laparoscopic abdominal surgery
* General anesthesia lasting 2 hours or longer.

Exclusion Criteria:

* 1. Planned postoperative mechanical ventilation
* 2. Planned regional anesthesia/analgesia
* 3. Perioperative gabapentin, magnesium, or nitrous oxide use
* 4. Pregnancy or breastfeeding
* 5. Morbid obesity (BMI ≥ 35 kg/m2)
* 6. American Society of Anesthesiologists (ASA) physical status IV-V
* 7. Allergy to study medications
* 8. Contraindication to lidocaine (severe cardiac arrhythmia)
* 9. Contraindication to ketamine (psychiatric disorder, substance abuse, uncontrolled hypertension, pulmonary hypertension, increased intracranial or intraocular pressure, use of monoamine oxidase inhibitors)
* 10. Chronic preoperative opioid use (≥ 90 morphine mg equivalents per day for > 3 months)
* 11. Significant preoperative hepatic dysfunction (alanine aminotransferase or aspartate aminotransferase levels > 5 times normal) or planned liver transplantation
* 12. Preoperative cardiac failure (left ventricular ejection fraction ≤ 40%)
* 13. Unable to communicate or comprehend study instructions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pain scores | First postoperative 48 hours (measured at the end of the PACU stay as well as on the 1st and 2nd postoperative mornings).
  Pain scores based on the visual analog scale and Brief Pain Inventory. Ranges from 0 to 10, with 0 being no pain and 10 being the worst imaginable pain. The intervention will be deemed effective if both outcomes are non-inferior, and at least one is superior, to the control group.
Total opioid consumption | First postoperative 48 hours
  Total opioid consumption in oral morphine equivalents (mg) from the time of transfer to PACU through to the second postoperative morning. The intervention will be deemed effective if both outcomes are non-inferior, and at least one is superior, to the control group.

SECONDARY OUTCOMES:
Overall benefit of analgesia score (OBAS) | First postoperative 48 hours (measured at the end of the PACU stay as well as on the 1st and 2nd postoperative mornings).
  Measures 7 different items, i.e. current pain, vomiting, itching, sweating, freezing, dizziness, and patient satisfaction related to pain management. Each item is scored from 0 to 4, with the total OBAS score ranging from 0 to 28. The lower the total OBAS score, the higher the benefit of analgesia.
Quality of recovery (QoR-15) score | First postoperative 48 hours (measured at the end of the PACU stay as well as on the 1st and 2nd postoperative mornings).
  Measures 15 different items, i.e. ability to breathe easily, enjoy food, feel rested, have a good sleep, look after personal toilet and hygiene unaided, communicate with family or friends, getting support from hospital doctors and nurses, return to work or usual home activities, feel comfortable and in control, have a feeling of general well-being, as well as the presence of moderate pain, severe pain, nausea or vomiting, feeling worried or anxious, and feeling sad or depressed. Each item is scored from 0 to 10, with a total QoR-15 score ranging from 0 to 150. The higher the QoR-15 score, the better the quality of recovery in the postoperative period.

OTHER OUTCOMES:
Time to first opioid administration | The amount of time from PACU admission to PACU discharge
  Measured in minutes
Postoperative hospital length of stay | The number of days from hospital admission to hospital discharge
  Measured in days
Nausea or vomiting | First postoperative 48 hours
  Measured as dichotomous outcome (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Minear, MD, Principal Investigator — Cleveland Clinic Florida
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grady MV, Mascha E, Sessler DI, Kurz A. The effect of perioperative intravenous lidocaine and ketamine on recovery after abdominal hysterectomy. Anesth Analg. 2012 Nov;115(5):1078-84. doi: 10.1213/ANE.0b013e3182662e01. Epub 2012 Sep 25. PMID 23011561
- [Background] Weibel S, Jelting Y, Pace NL, Helf A, Eberhart LH, Hahnenkamp K, Hollmann MW, Poepping DM, Schnabel A, Kranke P. Continuous intravenous perioperative lidocaine infusion for postoperative pain and recovery in adults. Cochrane Database Syst Rev. 2018 Jun 4;6(6):CD009642. doi: 10.1002/14651858.CD009642.pub3. PMID 29864216
- [Background] Elia N, Tramer MR. Ketamine and postoperative pain--a quantitative systematic review of randomised trials. Pain. 2005 Jan;113(1-2):61-70. doi: 10.1016/j.pain.2004.09.036. PMID 15621365
- [Background] Ye F, Wu Y, Zhou C. Effect of intravenous ketamine for postoperative analgesia in patients undergoing laparoscopic cholecystectomy: A meta-analysis. Medicine (Baltimore). 2017 Dec;96(51):e9147. doi: 10.1097/MD.0000000000009147. PMID 29390443
- [Background] Zhao JB, Li YL, Wang YM, Teng JL, Xia DY, Zhao JS, Li FL. Intravenous lidocaine infusion for pain control after laparoscopic cholecystectomy: A meta-analysis of randomized controlled trials. Medicine (Baltimore). 2018 Feb;97(5):e9771. doi: 10.1097/MD.0000000000009771. PMID 29384867
- [Background] Sun Y, Li T, Wang N, Yun Y, Gan TJ. Perioperative systemic lidocaine for postoperative analgesia and recovery after abdominal surgery: a meta-analysis of randomized controlled trials. Dis Colon Rectum. 2012 Nov;55(11):1183-94. doi: 10.1097/DCR.0b013e318259bcd8. PMID 23044681

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/48/NCT04084548/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/48/NCT04084548/ICF_001.pdf